CLINICAL TRIAL: NCT07224880
Title: Safety and Outcomes of Ellacor® Micro-Coring Technology® in Fitzpatrick Skin Types I-VI, Including Patients Receiving Glucagon-Like Peptide-1 Receptor Agonists (GLP-1 RAs): A Case Series
Brief Title: Ellacor® Micro-Coring Technology® in Fitzpatrick Skin Types I-VI, Including Patients Receiving Glucagon-Like Peptide-1 Receptor Agonists
Status: Recruiting | Type: Observational
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-00457
Record Dates: First submitted 2025-10-29; First posted 2025-11-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: glp1 Agonist; Gene Expression; Skin Laxity
Keywords: ellacor; GLP-1; weight loss
MeSH Terms: conditions — Cutis Laxa; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted cores may be retained in the tubing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GLP1 Patients: Patients have lost at least 10% of their baseline body weight from taking a GLP-1 receptor agonist
  Interventions: Device: ellacor

INTERVENTIONS:
Device: ellacor — dermal non-thermal micro-coring device
  Other Names: micro-coring; dermal micro-coring

SUMMARY:
The main purpose of the study is to collect information about how the device functions in a variety of treatment areas and skin types and to find out what changes, if any, occur in the skin treated with the study device compared to the skin that wasn't treated including patients receiving GLP-1's, a class of medications that mimic a natural hormone to help control blood sugar and support weight loss. The study will also evaluate side effects that occur with this treatment, if any. Standardized 2D Imaging will be used to quantify reduction of wrinkle severity

DETAILED DESCRIPTION:
This device has been approved for sale by the United States Food and Administration (FDA) for use in treatment of moderate and severe wrinkles in the mid and lower face. This device is not currently approved by the FDA for use in other locations or for other indications. The study device uses specially designed hollow coring needles, that when inserted in the tissue remove cores the size of the needle inner diameter. The tissue cores are then removed from the needle and pulled out by suction. Compared to micro-needling procedures that only puncture the skin without removing any tissue, the ellacor Micro-Coring procedure needle removes full thickness cores of skin with diameters in the range of 400 microns (0.4 millimeters or about 4 times as wide as a human hair). Skin that is removed with the ellacor Micro-Coring Technology is below the size limit that causes visible scar formation. After study treatment with the MicroCoring Technology, the areas undergo a process of repair including the formation of new collagen and elastin fibers that are typical of healthy tissue.

A minimum of 10 and maximum of 30 people will participate in this study at Tri Valley Plastic Surgery. Tri Valley Plastic Surgery is the only center participating in this study. Each person in this study will receive the same number of ellacor® treatments The study will last up to 3 months (90 days) for each person participating. There will be a minimum of 6 study visits: a Screening & Enrollment Visit followed by 1 ellacor treatment visit and 4 followup visits (Day 3, Day 7, Day 30, and Day 90); there may be an addition follow-up visit as needed according to you and your doctor. Each visit is estimated to take 30 to 90 minutes. Your participation in the study ends on the Day 90 follow-up visit. Your screening visit and your first ellacor treatment visit could occur on the same day. If this happens then your participation in the study will be about 3 months (90 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult, between the ages of 30 and 65
2. Fitzpatrick Skin Type I-VI
3. Have moderate to severe wrinkles on the mid and lower face, according to Lemperle Wrinkle Severity Scale (LWSS), i.e. score 3, 4 or 5.
4. Have moderate to extreme abdominal laxity according to Stokes Scale (i.e., score of 2-4 on a scale of 0-4).
5. Willingness to sign Informed Consent Form

Exclusion Criteria:

1. Pregnant women or nursing mothers
2. Patients with dermatosis, open wounds, sores, or irritated skin in the treatment area
3. Patients with allergy to stainless steel or to topical, oral, or injected medications or preparations that may be used during the procedure, such as petrolatum, lidocaine, bupivacaine, chlorhexidine, or povidone-iodine
4. Patients with a history or presence of any clinically significant bleeding disorder
5. Patients with dermatological or autoimmune conditions that may affect the treatment outcome; these may include, but are not limited to: actinic keratosis, raised nevi, rosacea, melasma, active acne, cutaneous papules/nodules, active inflammatory lesions, dermatitis, psoriasis, cellulitis, urticarial folliculitis, acute inflammatory phase of scleroderma, rheumatoid arthritis, eczema, psoriasis, allergic dermatitis, collagen disorders, or lupus
6. Patients with systemic infections or acute local skin infections (as Hepatitis disorders type A, B, C, D, E or F or HIV infection)
7. Patients who are on a high dose of anti-coagulants or blood-thinning substances, e.g., aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), warfarin, heparin, acetylsalicylic acid during the previous fourteen (14) days
8. Patients who are on courses of chemotherapy, high-dose corticosteroid use, or radiation in the treatment area
9. Patients with have undergone plastic surgery of the face within the last twelve (12) months or have any facial surgical scars less than twelve (12) months old
10. Patients who have undergone injections of dermal fillers, fat, or botulinum toxin, as well as any minimally invasive/invasive skin treatment in the treatment area during the previous six (6) months
11. Patients with scars less than six (6) months old in the treatment area

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult male and female participants aged between 30 to 65 years, with FST I-VI, with moderate to severe mid to lower face wrinkles and/or abdominal skin laxity as a result of excessive weight loss. They have chosen to participate in this study as evidenced by execution of the informed consent document.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and Outcomes | study time frame
  Safety and Efficacy of ellacor treatment in participants with FST I-VI, inclusive of participants following treatment with GLP-1 RA
  There will be follow-up appointments after the initial screening and enrollment visit. Each of the assessments at follow up days are specified below:
  Baseline or Day 0 Day 3 Day 7 Day 30 through study completion, up to Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Tri Valley Plastic Surgery, Dublin, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subedi SK, Ganor O. Considerations for the Use of Fitzpatrick Skin Type in Plastic Surgery Research. Plast Reconstr Surg Glob Open. 2024 Jun 5;12(6):e5866. doi: 10.1097/GOX.0000000000005866. eCollection 2024 Jun. No abstract available. PMID 38841534
- [Background] Gfrerer L, Kilmer SL, Waibel JS, Geronemus RG, Biesman BS. Dermal Micro-coring for the Treatment of Moderate to Severe Facial Wrinkles. Plast Reconstr Surg Glob Open. 2022 Oct 17;10(10):e4547. doi: 10.1097/GOX.0000000000004547. eCollection 2022 Oct. PMID 36262685